CLINICAL TRIAL: NCT05943301
Title: Study of the Impact of Non-pharmacological Techniques (Self-hypnosis/Self-care) on the Well-being, Cognitive Complaints and Return-to-work in Cancer Patients
Brief Title: Study of the Impact of Non-pharmacological Techniques on Cognitive Complaints in Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with recruitment
Sponsor: University of Liege (Other)
Collaborators: Fondation Benoit (Unknown)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, PhD, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/204
Record Dates: First submitted 2019-02-11; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Non-Metastatic Neoplasm
Keywords: Cancer; Hypnosis; Self-care; Cognition
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Each participant will be tested by the experimenter on T0. One month later, the experimenter will assess all participants (T1). After that, a person external from the study will randomize participants to the experimental group or the controle group. The experimental group will proceed to an 8 week (1 session of 2 hours a week) training programme of self-hypnosis/self-care with a therapist specialized in hypnosis, while the group control will be on waiting list. After this learning phase, all participant will be assessed once again (T2). Then, the group control will enter the learning phase. After the completion of this learning phase/waiting list, all participants will proceed to a last evaluation (T3) to assess the self-hypnosis/self-care effect over time.
Who Masked: Investigator
Masking Description: The investigator will not know which participant is in the learning phase or in the waiting list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Self-hypnosis/self-care intervention : It is an 8-week 2 hour-session (one session per week) of self-hypnosis/ self-care learning. Participants are given strategies to learn self-care (knowing your own needs, self-respect, communication, etc.), each strategie is discussed for participant to understand them and thus applie them correctly in daily living. An hypnosis exercice is also realised at the end of each session.
  Interventions: Behavioral: Self-hypnosis/self-care
- Control group (No Intervention): The control goup has usual care and no intervention.

INTERVENTIONS:
Behavioral: Self-hypnosis/self-care — Learning phase of self-hypnosis/self-care
  Arms: Experimental group

SUMMARY:
Cancer diagnosis generates a number of physical (pain, nausea and fatigue) and psychological implications for the patient. At the psychological level, there are high levels of emotional distress (anxiety and depression) and cognitive impairments such as memory, attentional and information processing deficits, that can undermine the quality of life. This last decade has shown great progress in cancer treatment allowing cancer patients, many of whom are of working age, to survive. Unfortunately, cancer diagnosis and treatment induce various symptoms necessitating the patient to interrupt or quit his occupational status. Hypnosis has been used in the past few years to treat these psychological and physical symptoms, be it at the moment of diagnosis, during and/or after the cancer treatments. A large amount of studies has shown a positive effect of hypnosis in cancer patients notably upon anxiety, emotional distress and fatigue, three factors that can negatively affect cognitive functions. The purpose of our study is to investigate the effect of a non-pharmacological treatment that combines self-hypnosis and self-care on well-being, cognitive complaints and return-to- work within a population of cancer patients. Our hypothesis is that, by reducing emotional distress and fatigue, self-hypnosis/self-care will reduce the cognitive difficulties of cancer patients, foster return-to-work, and eventually improve the patients' global quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Major
* Fluency in French
* End of surgery and/or chimiotherapy and/or radiotherapy : 1-12 months.
* Cognitive complaints

Exclusion Criteria:

* Brain cancer
* Metastatic cancer
* Psychiatric disorder
* Neurologic disorder
* Neuropsychological assessment made within 3 months
* Drug addiction
* Alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change in subjective cognitive difficulties : Perceived cognitive impairments | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on the perceived cognitive impairments will be assessed by means of the subtest "Perceived cognitive impairments" of the Functionnal Assessment of Cancer Therapy-Cognitive Function (FACT-COG; Wagner et al., 2009). Scale ranging from 0 to 4 (0=never; 4=several times a day).
Change in subjective cognitive difficulties : Comments by others | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on the perceived cognitive impairments will be assessed by means of the subtest "Comments by others" of the Functionnal Assessment of Cancer Therapy-Cognitive Function (FACT-COG; Wagner et al., 2009). Scale ranging from 0 to 4 (0=never; 4=several times a day).
Change in subjective cognitive difficulties : Perceived cognitive abilities | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on the perceived cognitive impairments will be assessed by means of the subtest "Perceived cognitive abilities" of the Functionnal Assessment of Cancer Therapy-Cognitive Function (FACT-COG; Wagner et al., 2009). Scale ranging from 0 to 4 (0=not at all; 4=very much).
Change in subjective cognitive difficulties : Impact on quality of life | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on the perceived cognitive impairments will be assessed by means of the subtest "Impact on quality of life" of the Functionnal Assessment of Cancer Therapy-Cognitive Function (FACT-COG; Wagner et al., 2009). Scale ranging from 0 to 4 (0=not at all; 4=very much).
Change in objective cognitive difficulties : Verbal long term memory | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on verbal long term memory will be assessed by means the Buschke Selective Reminding Test (Buschke, 1973). According to the sex and the subject's age, the test gives us a score and the norms.
Change in objective cognitive difficulties : Attention | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on attention abilities will be assessed by means of the subtest "Phasic alertness" of the Test of Attentional Performance 2.3.1 (Zimmermann & Fimm, 2002). Computerized test, according to the sex and the subject's age, the test gives us a score and the norms.
Change in objective cognitive difficulties : Processing speed | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on processing speed abilities will be assessed by means of the first part of the Stroop test (Stroop, 1935). According to the sex and the subject's age, the test gives us a score and the norms.
Change in objective cognitvie difficulties : Inhibition | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on inhibition abilities will be assessed by means of the first part of the Stroop test (Stroop, 1935). According to the sex and the subject's age, the test gives us a score and the norms.
Change in objective cognitvie difficulties : mental flexibility | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on mental flexibility abilities will be assessed by means of the subtest "Flexibility" of the Test of Attentional Performance 2.3.1 (Zimmermann & Fimm, 2002). Computerized test, according to the sex and the subject's age, the test gives us a score and the norms.
Change in objective cognitvie difficulties : working memory | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on mental flexibility abilities will be assessed by means of the subtest "Working memory" of the Test of Attentional Performance 2.3.1 (Zimmermann & Fimm, 2002). Computerized test, according to the sex and the subject's age, the test gives us a score and the norms.
Change in objective cognitvie difficulties : executive functions | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on executive functions will be assessed by means of the Wisconsin Card Sorting Test (David et al., 1948). According to the sex and the subject's age, the test gives us a score and the norms.
Impact on return-to-work | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  For people who continued to work at time of recruitment, Work Design questionnaire will be administered Morgeson & Hymphrey, 2006). Scale raging from 0 to 5 (0=not at all; 5=exactly).

SECONDARY OUTCOMES:
Change in emtional distress : Anxiety | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on anxiety and despression will be assessed by means of the Hopsital Anxiety and Depression Scale (Zigmond & Snaith, 1983). Scale ranging from 0 to 3 (0=never; 4=always).
Change in emtional distress : Depression | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on anxiety and despression will be assessed by means of the Hopsital Anxiety and Depression Scale (Zigmond & Snaith, 1983). Scale ranging from 0 to 3 (0=alwaysr; 4=never).
Change in fatigue : General fatigue | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on fatigue will be assessed by means of the subscale "general fatigue" of the Multidimensional Fatigue Inventory (Smets et al., 1995). Scale ranging from 1 to 4 (1=not agree at all; 4=agree completely).
Change in fatigue : Physical fatigue | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on fatigue will be assessed by means of the subscale "physical fatigue" of the Multidimensional Fatigue Inventory (Smets et al., 1995). Scale ranging from 1 to 4 (1=not agree at all; 4=agree completely).
Change in fatigue : Mental fatigue | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on fatigue will be assessed by means of the subscale "mental fatigue" of the Multidimensional Fatigue Inventory (Smets et al., 1995). Scale ranging from 1 to 4 (1=not agree at all; 4=agree completely).
Change in fatigue : Motivational decrease | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on fatigue will be assessed by means of the subscale "motivational decrease" of the Multidimensional Fatigue Inventory (Smets et al., 1995). Scale ranging from 1 to 4 (1=not agree at all; 4=agree completely).
Change in fatigue | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The impact of self-hypnosis/self-care on fatigue will be assessed by means of the Multidimensional Fatigue Inventory (MFI; Smets et al., 1995) and an 1-week agenda.
Change in fatigue : Weekly agenda | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  Qualitative questionnaire concerning the sleep habits of participants. They have to give information concerning their sleeping habits.
Change in quality of life | T1 (before the intervention), T2 (right after the intervention), T3 (3 months follow-up)
  The improvement of quality of life will be assessed my means of the european Organization for Reasearch and Treatment of Cancer QLQ-C30 version 3.0 (E Aaronson et al., 1993). Scale ranging from 1 to 4 (1=not at all; 4=excellent).

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - University of Liège, Liège
  - University, Liège

IPD SHARING:
Plan to Share IPD: No